CLINICAL TRIAL: NCT06255288
Title: A Nurse-led Intervention Consisting of a Structured Dialogue, Patient and Relative Information, and Protein Supplement for Patients with Leg Ulcers in Clinical Practice: a Feasibility Study
Brief Title: Time to Heal (Wound, Healing, Dialogue, Nutrition)
Acronym: SNAK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Roskilde University (Other)
Responsible Party: Principal Investigator, Pia Søe Jensen, Postdoc and Associate Professor, Hvidovre University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: F-23054461
Record Dates: First submitted 2024-01-25; First posted 2024-02-13 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-02

CONDITIONS: Leg Ulcer; Venous Leg Ulcer; Arterial Leg Ulcer; Foot Ulcer, Diabetic; Amputation Stump
Keywords: Leg ulcer; Nutrition; Dialogue; Diet; Nursing
MeSH Terms: conditions — Leg Ulcer; Varicose Ulcer; Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dialogue, patient information and protein supplement (Experimental): Patient will receive:
  1. Structured nutritional dialogue during two visits to the clinic.
  2. Written patient information (pamphlet) during their first visit to the clinic.
  3. Protein supplement drink during two visits to the clinic.
  4. Prescription of protein supplement drink during their first visit to the clinic.
  Interventions: Other: SNAK intervention

INTERVENTIONS:
Other: SNAK intervention — The intervention consists of structured dialogue, patient information, and a protein supplement. The structured dialogue part of the intervention consists of an A3 poster with illustrations and keywords which will be hanging in the outpatient clinics. The poster will be utilized by nurses, patients, and their relatives to facilitate a dialogue regarding nutrition and wound healing. The patient information part of the intervention consists of a leaflet with easy-to-read information, which patients and their relatives can bring home after their visit to the outpatient clinic. The leaflet will consist of general information as well as food categories and recipes they can use to enhance their daily protein intake. For the protein supplement part of the intervention, the patients will have access to protein supplement beverages while they are in the outpatient clinic waiting room. Furthermore, they will receive prescriptions for protein drinks, that they can pick up at their local pharmacy.

SUMMARY:
The objective of this study is to examine the feasibility, acceptability, fidelity, and outcome of a nurse-led nutritional intervention for patients with leg ulcers in a outpatient clinics. The intervention consists of a structured dialogue and patient information on key lifestyle behaviours to improve wound healing. Furthermore, the intervention includes protein supplement.

DETAILED DESCRIPTION:
The study aims to address the following research questions:

Primary Research Questions:

1. Is the patient recruitment process feasible?
2. Is the delivery of the intervention feasible?
3. Is the intervention acceptable to the patients?
4. Is the intervention acceptable to the nurses?
5. Is the intervention consistently maintained during the study period?
6. Are the data collection procedures feasible?
7. Are the outcome measures feasible?
8. What are the reasons for any dropouts?

Secondary Research Questions:

1. What are the patients' and relatives' views on receiving the intervention?
2. Are there any longitudinal differences in outcomes for the patient group?
3. Are there any individual patient-specific differences in outcomes over time?

The feasibility study will recruit patients with a first-time referral to the outpatient clinic at the Department of Orthopaedic Surgery at Copenhagen University Hospital, Hvidovre, for leg ulcers caused by arterial or venous disease or neuropathy due to diabetes. The intervention will be administered by the clinic's nurses.

After inclusion, each patient will be contacted by telephone following their next two clinic visits. The initial follow-up will assess patient characteristics, information about their wound using the Wound-Qol Questionnaire, and their perspective on receiving the intervention. The second and final follow-up will consist of an interview exploring their perspective on receiving the intervention. Additionally, focus group interviews with the nurses will be conducted to investigate their capability, opportunity, and motivation (COM-B model) for implementing the intervention. Both patient and nurse interviews will be recorded and transcribed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with leg ulcers caused by arterial or venous disease or neuropathy caused by diabetes.
* Patient with an amputation wound.
* Speak and understand Danish.

Exclusion Criteria:

* Patients with wounds caused by high-intensity trauma.
* Patients in the end-of-life phase.
* Patients living in nursing homes.
* Patients with cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
SNAK Feasibility questionnaire (SFQ) - Element 1: Evaluating structured dialogue | Measurements will be taken within 1 week after their second and third visits to the outpatient clinic. Each patient will be followed up to maximum 16 weeks after inclusion.
  The intervention is deemed non-feasible if, during their visit to the outpatient clinic, fewer than 80% of the patients:
  1. Noticed the dialogue tool.
  2. Had a conversation with the nurses about nutrition and wound healing using the dialogue tool.
  3. Found the conversation with the nurses about nutrition and wound healing relevant and valuable.
  4. Considered it acceptable to have a conversation with the nurses about nutrition and wound healing.
  The SFQ has two scoring systems: 1) Binary scores (yes/no) with a non-applicable option as well and 2) categorical 5-point score (1 is the highest score and 5 is the lowest score in regards to agreement on statements related to the interventions feasibility). The 5-point categorical score will be presented with median and interquartile ranges (IQR).
SNAK Feasibility questionnaire (SFQ) - Element 2: Evaluating patient and relative information | Measurements will be taken within 1 week after their second and third visits to the outpatient clinic. Each patient will be followed up to maximum 16 weeks after inclusion.
  The intervention is considered non-feasible if, during their visit to the outpatient clinic, fewer than 80% of the patients:
  1. Received a leaflet.
  2. Could read and understand the leaflet.
  3. Found the information in the leaflet relevant.
  4. have attempted to use the suggested recipes or food categories.
  5. have attempted to change their diet.
  The SFQ has two scoring systems: 1) Binary scores (yes/no) with a non-applicable option as well and 2) categorical 5-point score (1 is the highest score and 5 is the lowest score in regards to agreement on statements related to the interventions feasibility). The 5-point categorical score will be presented with median and interquartile ranges (IQR).
SNAK Feasibility questionnaire (SFQ) - Element 3: Evaluating protein supplement | Measurements will be taken within 1 week after their second and third visits to the outpatient clinic. Each patient will be followed up to maximum 16 weeks after inclusion.
  The intervention is considered non-feasible if, during their visit to the outpatient clinic, fewer than 80% of the patients:
  1. Were offered a protein supplement drink.
  2. Were offered a prescription for protein supplement drinks.
  3. Agree that patients should be offered a protein supplement drink.
  The SFQ has two scoring systems: 1) Binary scores (yes/no) with a non-applicable option as well and 2) categorical 5-point score (1 is the highest score and 5 is the lowest score in regards to agreement on statements related to the interventions feasibility). The 5-point categorical score will be presented with median and interquartile ranges (IQR).
SNAK Feasibility questionnaire (SFQ) - Element 4: Evaluating overall intervention | Measurements will be taken within 1 week after their second and third visits to the outpatient clinic. Each patient will be followed up to maximum 16 weeks after inclusion.
  The intervention is considered non-feasible if fewer than 80% of the patients, during their visit to the outpatient clinic, are confident that they can follow the advice regarding nutrition and lifestyle in their daily lives.
  The SFQ has two scoring systems: 1) Binary scores (yes/no) with a non-applicable option as well and 2) categorical 5-point score (1 is the highest score and 5 is the lowest score in regards to agreement on statements related to the interventions feasibility). The 5-point categorical score will be presented with median and interquartile ranges (IQR).
Qualitative evaluation of nurses' Capability, Opportunity, and Motivation (COM-B) to implement the intervention. | Measured 16 weeks after first inclusion.
  COM-B will be explored using a semi-structured focus group interview with the nurses and will be carried out in the outpatient clinic following the end of inclusion (16 weeks after first inclusion).
Procedural uncertainties - Number of patients willing to participate. | Measured 4, 8, 12, and 16 weeks after first inclusion.
  Following criteria are considered to evaluate the recruitment of participation in the intervention.
  1. If less than 30% are willing to participate in the intervention, then the intervention is considered non-feasible.
  2. If recruitment falls within the range of 30 to 80% modification will be considered.
  If 80% or more are recruited, the study is deemed feasible without modification.

SECONDARY OUTCOMES:
Recruitment rates | Every week until study completion (16 weeks after first inclusion).
  The number of eligible patients that agree to participate will be collected.
Drop out rates | Every week until study completion (16 weeks after first inclusion).
  The number of included patients that withdraw consent or drop out for other reasons will be collected. Furthermore, we will collect reasons for dropout.

CONTACTS AND LOCATIONS:
Overall Officials: Pia Søe Jensen, Principal Investigator — Hvidovre University Hospital, Copenhagen
Locations (1):
- Outpatient clinic at the Department of Orthopedic Surgery, Hvidovre University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No